CLINICAL TRIAL: NCT04574102
Title: Clinical Investigation of Omega Refractive Capsule, Model V in Combination With a Commercially Available, FDA Approved Monofocal or Toric Intraocular Lens
Brief Title: Clinical Investigation of Omega Refractive Capsule Model V With Use of an FDA Approved IOL
Acronym: ORCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omega Ophthalmics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Omega Refractive Capsule Mod V
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This study is a prospective, interventional, randomized, controlled, paired eye, subject-masked design.
  Subjects will be randomly assigned to which eye will receive the Omega Refractive capsule V with an FDA approved intraocular lens. Fellow eyes will serve as controls and receive an FDA approved IOL (no Omega capsule).
Who Masked: Participant
Masking Description: subjects will be masked to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Eye (Experimental): Omega Refractive capsule, model V, with an FDA approved intraocular lens.
  Interventions: Device: Omega Refractive Capsule with FDA approved Intraocular Lens
- Control Eye (Active Comparator): FDA approved Intraocular Lens
  Interventions: Device: FDA approved Intraocular lens

INTERVENTIONS:
Device: Omega Refractive Capsule with FDA approved Intraocular Lens — Omega Refractive Capsule with FDA approved Intraocular Lens
  Other Names: FDA approved intraocular lens
  Arms: Study Eye
Device: FDA approved Intraocular lens — FDA approved Intraocular lens
  Arms: Control Eye

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the

investigational Omega Refractive Capsule (model V)

DETAILED DESCRIPTION:
This study is a prospective, interventional, randomized, controlled, paired eye, subject-masked design.

Subjects will be randomly assigned to which eye will receive the Omega Refractive capsule V with an FDA approved intraocular lens. Fellow eyes will serve as controls and receive an FDA approved IOL (no Omega capsule).

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older at the time of surgery diagnosed with bilateral cataracts
* Able to understand and sign an informed consent
* Willing and able to complete all study visits and assessments required for the study
* Calculated lens power within the available range
* Corrected distance visual acuity is equal to or worse than 20/40 in each eye with or without a glare source present
* Bilateral cataracts eligible for extraction by phacoemulsification and capsular bag fixated IOL implantation
* Potential postop visual acuity of 20/25 or better in the judgment of the surgeon
* Preoperative corneal astigmatism of 4.0 D or less with normal corneal topography
* Clear intraocular media other than cataract
* Preop endothelial cell density of 2000 cells/mm2 or more

Exclusion Criteria:

* Subject's best corrected vision is light perception or no light perception in either eye
* Cataract opacification preventing adequate Binocular Indirect Ophthalmoscopic retinal and macular examination.
* Orbital abnormalities, such as thyroid related orbitopathy, causing significant exophthalmos.
* Eyelid abnormalities causing lagophthalmos.
* Significant anterior blepharitis or meibomian gland dysfunction
* Corneal abnormalities or conditions, other than regular topographic corneal astigmatism
* Krukenburg's spindle (linear pigmentary deposits on the corneal endothelium)
* Abnormalities of the iris including trans-illumination defects
* Pupil abnormalities (abnormally shaped, fixed or non-reactive)
* Pharmacologic dilation less than 7 mm
* Axial length <22.5mm
* Lens thickness <4.1 mm
* Anterior chamber depth <2.5mm
* Prior ocular surgery
* Epiretinal membrane
* Macular edema
* Retinal tears including operculated holes
* Amblyopia
* Glaucoma of any kind
* Pseudoexfoliation syndrome
* History of uveitis/iritis
* Diabetic retinopathy
* Acute, chronic or uncontrolled systemic or ocular disease that may confound the results of the study (including rheumatologic conditions such as Rheumatoid arthritis, ankylosing spondyliltis, Sjögren's syndrome, and neurologic conditions such as optic neuritis or multiple sclerosis).
* Prior or anticipated use of tamsulosin or silodosin (e.g., Flomax®, Flomaxtra®, Rapaflo®) or similar medications
* Average Keratometry <38D or > 48D by topography
* Any pathology of the zonules including evidence of zonular weakness, zonular instability, zonular damage, or coloboma effecting zonules.
* History of ocular trauma
* Pregnant, lactating, or has another condition with associated fluctuation of hormones that could lead to refractive changes

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Absence of fusion of peripheral anterior and posterior capsule | 6 Month Postoperative Visit
  slit lamp exam

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Orlich, MD, Principal Investigator
Locations (1):
- Clinica 20/20, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No